CLINICAL TRIAL: NCT01200745
Title: Efficacy of Topical Capsaicin on Chronic Neck Pain ; Double-blinded Randomized Trial
Brief Title: Efficacy of Topical Capsaicin on Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Mi-Yeon Song / Department of Oriental Rehabilitation Medicine, College of Oriental Medicine, Kyung Hee University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHU 20100675
Record Dates: First submitted 2010-09-02; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Neck Pain
Keywords: neck pain; capsaicin; dermal patch
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- capsaicin patch (Active Comparator)
  Interventions: Drug: Capsaicin patch
- Hydrogel patch (Placebo Comparator)
  Interventions: Drug: Capsaicin patch

INTERVENTIONS:
Drug: Capsaicin patch — Over an four-week period, the treatment group (n=30) uses capsaicin patch (100 mcg/3cc) at the tender point of neck for 12 hours a day; the control group (n=30) receives Hydrogel patch instead of capsaicin patch.
  Other Names: Hydrogel Patch

SUMMARY:
The purpose of this study is to determine whether topical capsaicin patch can effectively reduce chronic neck pain.

DETAILED DESCRIPTION:
* Design: This is a double-blind, randomized, controlled study. Participants: Sixty participants with chronic neck pain are recruited and randomly assigned to two groups.
* Intervention: Over an four-week period, the treatment group (n=30) uses capsaicin patch (100 mcg/3cc) at the tender point of neck for 12 hours a day; the control group (n=30) receives Hydrogel patch instead of capsaicin patch.

ELIGIBILITY:
Inclusion Criteria:

* Korean participants with Chronic neck pain are enrolled in our study

Exclusion Criteria:

* Participants with coagulation deficiencies, infections, hypertension, diabetes, heart disease, renal disease, liver disease, cancer, myelopathy, hypersensitivity of drugs, other skeletomuscular disease, allergic response to capsaicin, pregnancy and nursing are excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analogue Scale(VAS) | 4 week

SECONDARY OUTCOMES:
Neck disability index | 4 week
  Neck disability index : questionnaire for measuring how much neck pain affects ability of daily activities
Beck depression inventory | 4 week
  Beck depression inventory : for assessing depression
SF-36 | 4 week
  questionnaire for measuring health-related quality of life
EQ-5D(EuroQol-5 dimension) | 4 week
  questionnaire for measuring health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Yeon Song, OMD, PhD, Principal Investigator — Department of Oriental Rehabilitation Medicine/College of Oriental Medicine/Kyung Hee University
Locations (1):
- Kyunghee University East West Neo Medical Center, Seoul, South Korea